CLINICAL TRIAL: NCT02764632
Title: Digital Facilitation of Nasogastric Tube Insertion Under General Anethesia
Brief Title: Facilitation of NGT Insertion
Acronym: NGT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, DR, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RefaNGT
Record Dates: First submitted 2016-05-05; First posted 2016-05-06 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Nasogasrtic Tube Insertion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Didgital group (Active Comparator): After induction of anesthesia, and after ensuring muscle relaxation, NGT will be inserted through the selected nostril and advanced for 12 cm then the NGT was advanced according to study group advancing. In control group; NGT was inserted with patient head flexed. In D group, after feeling the NGT in pharynx, with the head in neutral position,the index finger was used to support the NGT with slight direction towards the left side. This will prevent tube kinking at this point in front of the resistance offered by the inflated tube cuff or arytenoids cartilage. Also, this digital support reinforces the tube at the area weakened by its openings
  Interventions: Procedure: Digital facilitation
- Control group (No Intervention)

INTERVENTIONS:
Procedure: Digital facilitation
  Arms: Didgital group

SUMMARY:
Insertion of a nasogastric tube (NGT) in anesthetized patients can be a disappointing experience. Many techniques have been explained to improve success rate along with increasing safety, such as forward displacement of the larynx, tube rigidity improvement methods, pushing it down directly through pharynx or using a guide tube. Failure of insertion under general anesthesia reached 50% in some publications

ELIGIBILITY:
Inclusion Criteria:

* all surgicl patients needing NGT insertion

Exclusion Criteria:

* refusal coagulopathy ASA more than 2

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
NGT insertion success rate | intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dkahleya, Egypt

IPD SHARING:
Plan to Share IPD: Yes